CLINICAL TRIAL: NCT02950480
Title: Breast Capsular Contracture Following Post-Mastectomy Reconstruction in Women Treated With the Leukotriene Inhibitor Zafirlukast: A Phase II Trial
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15754
Record Dates: First submitted 2016-09-07; First posted 2016-11-01 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer
Keywords: Mastectomy
MeSH Terms: conditions — Breast Neoplasms | interventions — zafirlukast; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Zafirlukast (Experimental): Zafirlukast
  Interventions: Drug: zafirlukast
- Standard of Care (no intervention) (Other): Standard of Care (no intervention)
  Interventions: Other: Standard of Care (no intervention)

INTERVENTIONS:
Drug: zafirlukast — Patients will begin treatment with zafirlukast on post-operative day one following placement of tissue expander(s) once determined safe from a surgical recovery standpoint. They will be continued on the standard dosing (20mg PO twice per day) of zafirlukast through expander fill (6-12 weeks, up to 18 weeks for women receiving radiation). Treatment will be stopped 48 hours prior to expander-implant exchange, which is equivalent to five half-lives of the drug. Patients will be seen every 1 to 2 weeks for expander fill, and will be assessed clinically based on the Baker classification system of capsular contracture every two weeks.
  Other Names: Accolate
  Arms: Zafirlukast
Other: Standard of Care (no intervention) — Standard of Care (no intervention)
  Arms: Standard of Care (no intervention)

SUMMARY:
A 2 arm, 90 patient (45 per cohort) trial in patients with breast cancer who will be undergoing mastectomy with immediate tissue-expander reconstruction to determine whether treatment with zafirlukast (20mg PO BID) can reduce or prevent the development of capsular contracture.

DETAILED DESCRIPTION:
A 2 arm, 90 patient (45 per cohort) trial in patients with breast cancer who will be undergoing mastectomy with immediate tissue-expander reconstruction to determine whether treatment with zafirlukast (20mg PO BID) can reduce or prevent the development of capsular contracture.

Patients will be block randomized 1:1 into two cohorts: treatment with zafirlukast and the standard of care, or standard of care alone. Patients will begin treatment with zafirlukast on post-operative day one following placement of tissue expander(s) once determined safe from a surgical recovery standpoint. They will be continued on the standard dosing (20mg PO twice per day) of zafirlukast through expander fill (6-12 weeks, up to 18 weeks for women receiving radiation). Treatment will be stopped 48 hours prior to expander-implant exchange, which is equivalent to 5 half-lives of the drug. Patients will be seen every 1-2 weeks for expander fill, and will be assessed clinically based on the Baker classification system of capsular contracture at every appointment. The day of surgery for their expander-implant exchange, their Baker classification will also be noted.

During expander-implant exchange, three representative sections of the expander capsule will be collected: medial, lateral and anterior capsule specimens. These specimens will be bisected; half will be sent to pathology and half will be collected by the Munster lab. Gross and microscopic determination of capsule thickness will be performed by the pathology department. The Munster lab will fix and stain the tissues to look for the presence of collagen, level of fibrosis and number of myofibroblasts. Fibrosis level and collagen presence will be determined by performing immunohistochemistry with a Trichrome stain of the tissues, as well as Western blot analysis with Collagen-1. Myofibroblasts will be detected using immunohistochemistry with commercially available antibodies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are scheduled to undergo therapeutic or prophylactic mastectomy with immediate placement of tissue expanders and have a strong family history or hereditary cancer
2. Age ≥ 18 years
3. Zafirlukast is pregnancy category B. There are no adequate and well-controlled trials in pregnant women. Therefore, the effects of zafirlukast on the developing human fetus are unknown. For this reason, women of child-bearing potential must agree to use adequate contraception: 2 methods of birth control, prior to study entry ad for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.
4. Ability to understand a written informed consent document, and the willingness to sign it
5. At least 4 weeks post-completion of chemotherapy
6. Adequate organ function within 14 days start of study start:

   1. Absolute neutrophil count (ANC) ≥ 1.5 X 10^9/L
   2. Hemoglobin (Hgb) ≥9g/dL
   3. Platelets (plt) ≥ 100 x 10^9/L
   4. Potassium within normal range, or correctable with supplements;
   5. AST and ALT ≤2.5 x Upper Limit Normal (ULN) or ≤5.0 x ULN if liver tumor is present;
   6. Serum total bilirubin ≤ 1.5 x ULN
   7. Serum creatinine ≤ 1.5 x ULN, or 24-hr clearance ≥ 60ml/min

Exclusion Criteria:

1. Any significant medical condition, laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study
2. Currently on a leukotriene inhibitor or used within the past 6 months
3. Prior chest wall radiation
4. Pregnant or breastfeeding
5. Hepatic impairment as defined by:

   • AST(SGOT) > 2.5X institutional ULN and ALT(SGPT) > 2.5X institutional ULN
6. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela N Munster, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zafirlukast | Standard of Care (no Intervention)
Started | 2 | 2
Completed | 1 | 2
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zafirlukast | Standard of Care (no Intervention) | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Customized [Count of Participants; unit: Participants]
  30-39 | 0 | 1 | 1
  40-49 | 1 | 0 | 1
  50-59 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Capsular Thickness
Description: Compare capsular thickness by gross and microscopic measurement at the time of expander-implant exchange in those treated with zafirlukast (20 mg PO BID) compared with standard of care.
Time Frame: Day 44 to Day 126
Population: No participants were analyzed due to a change in post-mastectomy reconstruction standard practice which implements pre-pectoral implants resulting in low accruals to the protocol. The study was closed prior to any measurements taken or histology analyzed as there would have been insufficient data to produce any statistically significant results.
Arm/Group | Zafirlukast | Standard of Care (no Intervention)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Histologic Analysis: Compare Capsular Thickness by Gross and Microscopic Measurement at the Time of Expander-implant Exchange in Those Treated With Zafirlukast (20 mg PO BID) Compared With Standard of Care
Description: Perform histologic analysis of the capsule specimens to compare overall fibrosis and collagen deposition between the zafirlukast and standard of care groups.
  During expander-implant exchange, three representative sections of the expander capsule will be collected: medial, lateral and anterior capsule specimens. Gross and microscopic determination of capsule thickness will be performed by the pathology department. The Munster lab will fix and stain the tissues to look for the presence of collagen, level of fibrosis, and number of myofibroblasts. Fibrosis level and collagen presence will be determined by performing immunohistochemistry with a Trichrome stain of the tissues, as well as Western blot analysis with Collagen-1. Myofibroblasts will be detected using immunohistochemistry with commercially available antibodies.
Time Frame: Day 44 to Day 126
Population: as for outcome 1
Arm/Group | Zafirlukast | Standard of Care (no Intervention)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Appearance of Capsular Contracture
Description: The capsule tissue that is removed at the time of expander-implant exchange will be fixed and histologically assessed for the presence of fibroblasts and myofibroblasts.
Time Frame: After Day 44 to Day 126
Population: as for outcome 1
Arm/Group | Zafirlukast | Standard of Care (no Intervention)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events will be assessed at time of mastectomy and tissue expander placement (week 0), week 2, week 5, week 11, and week 17 until 30 days after treatment termination. Serious adverse events were collected for 30 days after the end of treatment, or until death, whichever occurs first. Patients removed from treatment for unacceptable treatment related adverse event(s) were followed until resolution or stabilization of all treatment related adverse events to Grade 1 or baseline.
Arm/Group | Zafirlukast | Standard of Care (no Intervention)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/2
Other Adverse Events (participants affected / at risk) | 1/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zafirlukast (N=2) | Standard of Care (no Intervention) (N=2)
Breast Infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zafirlukast (N=2) | Standard of Care (no Intervention) (N=2)
Fatigue (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 2 (2)
Edema limbs (General disorders) | 0 (0) | 1 (1)
Edema trunk (General disorders) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/80/NCT02950480/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/80/NCT02950480/Prot_SAP_001.pdf